CLINICAL TRIAL: NCT03554668
Title: The Relation Between Acute Changes in the Systemic Inflammatory Response, Thiamine and Magnesium Concentrations and Transketolase Activity After Elective Knee Arthroplasty.
Brief Title: Systemic Inflammatory Response: Thiamine and Magnesium Status (Sir TaM Study)
Acronym: SirTaM
Status: Completed | Type: Observational
Sponsor: Glasgow Royal Infirmary (Other)
Collaborators: NHS Greater Glasgow and Clyde (Other)
Responsible Party: Principal Investigator, Dr. Donogh Maguire, Emergency Medicine Clinical Researcher, Glasgow Royal Infirmary
Other Study IDs: REC reference 17/EE/0270; 225557 (Registry Identifier: IRAS)
Record Dates: First submitted 2018-05-31; First posted 2018-06-13 (Actual); Last update posted 2020-04-28 (Actual); Status verified 2020-04

CONDITIONS: Inflammation; Magnesium Deficiency; Iron-deficiency; Thiamine Deficiency
MeSH Terms: conditions — Inflammation; Magnesium Deficiency; Anemia, Iron-Deficiency; Thiamine Deficiency | interventions — Blood Specimen Collection

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Blood
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- 1: Post total knee replacement patients
  Interventions: Diagnostic Test: Blood draw

INTERVENTIONS:
Diagnostic Test: Blood draw — We take blood samples at pre-op and subsequent time points, up to three months post op.

SUMMARY:
We wish to determine to what extent magnesium, thiamine and transketolase activity are affected by the Systemic Inflammatory Response (SIR). The knee arthroplasty model affords the ideal study design, as surgery generates an inflammatory response.

Blood samples are drawn preoperatively and for up to four days post operatively, and again at three months post-operation.

DETAILED DESCRIPTION:
Thiamine and magnesium play a critical role in glucose metabolism and deficiency results in the accumulation of anaerobic metabolites including lactate (1-3).

Thiamine requires magnesium to be converted to its active form, thiamine pyrophosphate (TPP) (4). TPP also requires magnesium to achieve activation of TPP dependent enzymes during metabolism of glucose (5, 6). The 'gold standard' for the measurement of thiamine status is the measurement of Erythrocyte Transketolase Activity (ETKA)(4, 7-9), and this enzyme's activity is dependent on the presence both thiamine pyrophosphate and magnesium (8, 10). ETKA may therefore represent a 'functional marker' of magnesium status (7, 9, 11, 12).

Studies indicate that low plasma thiamine and magnesium are associated with a range of disease processes, many of which are inflammatory (13-17). Other lipid-soluble vitamins and minerals are known to decrease during the systemic inflammatory response (18, 19), however this relationship is not proven for magnesium. The systemic inflammatory response may therefore confound the interpretation of plasma thiamine and magnesium in the context of sepsis, surgery or autoimmune disease. Elective knee arthroplasty, provokes an inflammatory response and therefore provides an excellent controlled model for understanding the body's response to a systemic insult (19).

Obesity is reported to be associated with magnesium deficiency (17, 20). Intracellular magnesium plays a key role in regulating insulin action, insulin-mediated-glucose-uptake and vascular tone (21-23). Several epidemiologic studies have shown that adults and children consuming a western type diet are consuming 30 - 50% of the RDA for magnesium (24, 25). This deficiency appears to be predominantly subclinical and therefore not routinely investigated.

Obesity is also associated with thiamine and magnesium depletion (17, 20, 26, 27). Magnesium deficiency is also associated with a CRP rise (28-30). Thiamine status is proven to affect lactate concentrations in the blood (2, 3). Lactate accumulation is known to precede the onset of insulin resistance and be characteristically found in patients with obesity related diabetes (31-37).

It is therefore possible that an underlying quiescent magnesium and / or thiamine deficiency may mediate insulin resistance. Thiamine, and its more lipid soluble derivative, benfothiamine, have already shown some promise in the treatment of diabetic complications. The therapeutic potential is intriguing, however the relation between acute changes in the systemic inflammatory response and thiamine and magnesium concentrations, require clarification. Failure to prove the reliability of the thiamine and magnesium measurements in the context of the systemic inflammatory response may lead to patients receiving treatment for a measured deficiency of red cell thiamine and serum magnesium concentrations, which is unreliable. If the therapeutic potential of combined treatment with thiamine and magnesium for the optimization of ETKA function is to be realized (8), it is essential that the erythrocyte and plasma values used to determine thiamine status are definitively established in the context of the systemic inflammatory response. The knee arthroplasty model affords the ideal study design for this as there is a strong association between obesity and knee osteoarthritis (38, 39).

1. Andersen LW, Mackenhauer J, Roberts JC, Berg KM, Cocchi MN, Donnino MW. Etiology and therapeutic approach to elevated lactate levels. Mayo Clin Proc. 2013;88(10):1127-40.
2. Andersen LW, Holmberg MJ, Berg KM, Chase M, Cocchi MN, Sulmonte C, et al. Thiamine as an adjunctive therapy in cardiac surgery: a randomized, double-blind, placebo-controlled, phase II trial. Crit Care. 2016;20:92.
3. Moskowitz A, Lee J, Donnino MW, Mark R, Celi LA, Danziger J. The Association Between Admission Magnesium Concentrations and Lactic Acidosis in Critical Illness. J Intensive Care Med. 2016;31(3):187-92.
4. Lonsdale D. Thiamine and magnesium deficiencies: keys to disease. Med Hypotheses. 2015;84(2):129-34.
5. Lonsdale D. Thiamin(e): the spark of life. Subcell Biochem. 2012;56:199-227.
6. Bettendorff L, Wins P. Thiamin diphosphate in biological chemistry: new aspects of thiamin metabolism, especially triphosphate derivatives acting other than as cofactors. FEBS J. 2009;276(11):2917-25.
7. Kochetov GA, Solovjeva ON. Structure and functioning mechanism of transketolase. Biochim Biophys Acta. 2014;1844(9):1608-18.
8. Peake RW, Godber IM, Maguire D. The effect of magnesium administration on erythrocyte transketolase activity in alcoholic patients treated with thiamine. Scott Med J. 2013;58(3):139-42.
9. Sevostyanova IA, Yurshev VA, Solovjeva ON, Zabrodskaya SV, Kochetov GA. Effect of bivalent cations on the interaction of transketolase with its donor substrate. Proteins. 2008;71(2):541-5.
10. Dingwall KM, Delima JF, Gent D, Batey RG. Hypomagnesaemia and its potential impact on thiamine utilisation in patients with alcohol misuse at the Alice Springs Hospital. Drug Alcohol Rev. 2015;34(3):323-8.
11. Kochetov GA, Sevostyanova IA. Functional nonequivalence of transketolase active centers. IUBMB Life. 2010;62(11):797-802.
12. Meshalkina LE, Solovjeva ON, Khodak YA, Drutsa VL, Kochetov GA. Isolation and properties of human transketolase. Biochemistry (Mosc). 2010;75(7):873-80.
13. Liu D, Ke Z, Luo J. Thiamine Deficiency and Neurodegeneration: the Interplay Among Oxidative Stress, Endoplasmic Reticulum Stress, and Autophagy. Mol Neurobiol. 2016.
14. Georgiopoulos G, Chrysohoou C, Vogiatzi G, Magkas N, Bournelis I, Bampali S, et al. Vitamins in Heart Failure: Friend or Enemy? Curr Pharm Des. 2017.
15. Luong KV, Nguyen LT. The impact of thiamine treatment in the diabetes mellitus. J Clin Med Res. 2012;4(3):153-60.
16. Lima LF, Leite HP, Taddei JA. Low blood thiamine concentrations in children upon admission to the intensive care unit: risk factors and prognostic significance. Am J Clin Nutr. 2011;93(1):57-61.
17. Nielsen FH. Magnesium, inflammation, and obesity in chronic disease. Nutr Rev. 2010;68(6):333-40.
18. Ghashut RA, McMillan DC, Kinsella J, Talwar D. Erythrocyte concentrations of B1, B2, B6 but not plasma C and E are reliable indicators of nutrition status in the presence of systemic inflammation. Clin Nutr ESPEN. 2017;17:54-62.
19. Gray A, McMillan DC, Wilson C, Williamson C, O'Reilly DS, Talwar D. The relationship between the acute changes in the systemic inflammatory response, lipid soluble antioxidant vitamins and lipid peroxidation following elective knee arthroplasty. Clin Nutr. 2005;24(5):746-50.
20. Kerns JC, Arundel C, Chawla LS. Thiamin deficiency in people with obesity. Adv Nutr. 2015;6(2):147-53.
21. Barbagallo M, Dominguez LJ. Magnesium and type 2 diabetes. World J Diabetes. 2015;6(10):1152-7.
22. Mastrototaro L, Tietjen U, Sponder G, Vormann J, Aschenbach JR, Kolisek M. Insulin Modulates the Na+/Mg2+ Exchanger SLC41A1 and Influences Mg2+ Efflux from Intracellular Stores in Transgenic HEK293 Cells. J Nutr. 2015;145(11):2440-7.
23. Voma C, Etwebi Z, Soltani DA, Croniger C, Romani A. Low Hepatic Mg(2+) Content promotes Liver dysmetabolism: Implications for the Metabolic Syndrome. J Metab Syndr. 2014;3(4).
24. NHANES. What We Eat in America , NHANES 2013-2014, individuals 2 years and over (excluding breast-fed children) AveragThiamine and Magnesium https://www.ars.usda.gov/ARSUserFiles/80400530/pdf/1314/Table_1_NIN_GEN_13.pdf: www.ars.usda.gov/nea/bhnrc/fsrg. ; 2013 - 2014 [Average daily consumption of Thiamine and Magnesium 2013-4].
25. Altura BM, Shah NC, Shah GJ, Zhang A, Li W, Zheng T, et al. Short-term Mg deficiency upregulates protein kinase C isoforms in cardiovascular tissues and cells; relation to NF-kB, cytokines, ceramide salvage sphingolipid pathway and PKC-zeta: hypothesis and review. Int J Clin Exp Med. 2014;7(1):1-21.
26. Wolf E, Utech M, Stehle P, Büsing M, Stoffel-Wagner B, Ellinger S. Preoperative micronutrient status in morbidly obese patients before undergoing bariatric surgery: results of a cross-sectional study. Surg Obes Relat Dis. 2015;11(5):1157-63.
27. Farhanghi MA, Mahboob S, Ostadrahimi A. Obesity induced magnesium deficiency can be treated by vitamin D supplementation. J Pak Med Assoc. 2009;59(4):258-61.
28. Welch AA, Kelaiditi E, Jennings A, Steves CJ, Spector TD, MacGregor A. Dietary Magnesium Is Positively Associated With Skeletal Muscle Power and Indices of Muscle Mass and May Attenuate the Association Between Circulating C-Reactive Protein and Muscle Mass in Women. J Bone Miner Res. 2016;31(2):317-25.
29. Zuza EP, Barroso EM, Fabricio M, Carrareto AL, Toledo BE, J RP. Lipid profile and high-sensitivity C-reactive protein levels in obese and non-obese subjects undergoing non-surgical periodontal therapy. J Oral Sci. 2016;58(3):423-30.
30. Dibaba DT, Xun P, He K. Dietary magnesium intake is inversely associated with serum C-reactive protein levels: meta-analysis and systematic review. Eur J Clin Nutr. 2014;68(4):510-6.
31. Crawford SO, Hoogeveen RC, Brancati FL, Astor BC, Ballantyne CM, Schmidt MI, et al. Association of blood lactate with type 2 diabetes: the Atherosclerosis Risk in Communities Carotid MRI Study. Int J Epidemiol. 2010;39(6):1647-55.
32. Qvisth V, Hagström-Toft E, Moberg E, Sjöberg S, Bolinder J. Lactate release from adipose tissue and skeletal muscle in vivo: defective insulin regulation in insulin-resistant obese women. Am J Physiol Endocrinol Metab. 2007;292(3):E709-14.
33. Jansson PA, Larsson A, Smith U, Lönnroth P. Lactate release from the subcutaneous tissue in lean and obese men. J Clin Invest. 1994;93(1):240-6.
34. Chen YD, Varasteh BB, Reaven GM. Plasma lactate concentration in obesity and type 2 diabetes. Diabete Metab. 1993;19(4):348-54.
35. Lovejoy J, Newby FD, Gebhart SS, DiGirolamo M. Insulin resistance in obesity is associated with elevated basal lactate levels and diminished lactate appearance following intravenous glucose and insulin. Metabolism. 1992;41(1):22-7.
36. Lovejoy J, Mellen B, Digirolamo M. Lactate generation following glucose ingestion: relation to obesity, carbohydrate tolerance and insulin sensitivity. Int J Obes. 1990;14(10):843-55.
37. Kreisberg RA, Pennington LF, Boshell BR. Lactate turnover and gluconeogenesis in obesity. Effect of phenformin. Diabetes. 1970;19(1):64-9.
38. Guenther D, Schmidl S, Klatte TO, Widhalm HK, Omar M, Krettek C, et al. Overweight and obesity in hip and knee arthroplasty: Evaluation of 6078 cases. World J Orthop. 2015;6(1):137-44.
39. Salih S, Sutton P. Obesity, knee osteoarthritis and knee arthroplasty: a review. BMC Sports Sci Med Rehabil. 2013;5(1):25.

ELIGIBILITY:
Inclusion Criteria:

* undergoing elective total knee replacement

Exclusion Criteria:

* taking multivitamin

Ages: 18 Years to 99 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Patients undergoing elective TKR
Sampling Method: Non-Probability Sample
Enrollment: 47 (Actual)
Dates: Start 2018-01-15 (Actual); Primary Completion 2019-06-01 (Actual); Study Completion 2019-06-01 (Actual)

PRIMARY OUTCOMES:
serum magnesium | three months
  blood sample
thiamine | three months
  blood sample
erythrocyte transketolase activity | three months
  blood sample

OTHER OUTCOMES:
Iron receptor status | three months
  blood sample

CONTACTS AND LOCATIONS:
Locations (1):
- Glasgow Royal Infirmary, Glasgow, United Kingdom

IPD SHARING:
Plan to Share IPD: No
We will publish anonymised results. No patient identifiable data will be shared.

REFERENCES:
- [Background] Altura BM, Shah NC, Shah GJ, Zhang A, Li W, Zheng T, Perez-Albela JL, Altura BT. Short-term Mg deficiency upregulates protein kinase C isoforms in cardiovascular tissues and cells; relation to NF-kB, cytokines, ceramide salvage sphingolipid pathway and PKC-zeta: hypothesis and review. Int J Clin Exp Med. 2014 Jan 15;7(1):1-21. eCollection 2014. PMID 24482684
- [Background] Wolf E, Utech M, Stehle P, Busing M, Stoffel-Wagner B, Ellinger S. Preoperative micronutrient status in morbidly obese patients before undergoing bariatric surgery: results of a cross-sectional study. Surg Obes Relat Dis. 2015 Sep-Oct;11(5):1157-63. doi: 10.1016/j.soard.2015.03.018. Epub 2015 Apr 2. PMID 25980331
- [Background] Dibaba DT, Xun P, He K. Dietary magnesium intake is inversely associated with serum C-reactive protein levels: meta-analysis and systematic review. Eur J Clin Nutr. 2015 Mar;69(3):409. doi: 10.1038/ejcn.2014.275. Epub 2015 Jan 7. No abstract available. PMID 25563736
- [Background] Crawford SO, Hoogeveen RC, Brancati FL, Astor BC, Ballantyne CM, Schmidt MI, Young JH. Association of blood lactate with type 2 diabetes: the Atherosclerosis Risk in Communities Carotid MRI Study. Int J Epidemiol. 2010 Dec;39(6):1647-55. doi: 10.1093/ije/dyq126. Epub 2010 Aug 25. PMID 20797988
- [Background] Salih S, Sutton P. Obesity, knee osteoarthritis and knee arthroplasty: a review. BMC Sports Sci Med Rehabil. 2013 Dec 4;5(1):25. doi: 10.1186/2052-1847-5-25. PMID 24304704
- [Derived] Maguire D, Catchpole A, Sheerins O, Talwar D, Burns A, Blyth M, Shaw A, Jones B, Drury C, Harten J, Smith I, McMillan DC. The relation between acute changes in the systemic inflammatory response and circulating thiamine and magnesium concentrations after elective knee arthroplasty. Sci Rep. 2021 May 28;11(1):11271. doi: 10.1038/s41598-021-90591-y. PMID 34050237
- See also: What we eat in America - Magnesium deficiency — https://www.ars.usda.gov/ARSUserFiles/80400530/pdf/1314/Table_1_NIN_GEN_13.pdf